CLINICAL TRIAL: NCT05259020
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Cross-over, Clinical Trial to Evaluate the Pharmacokinetics and the Safety of ID14009 Compared to Coadministration of ID1805 With ID1803 in Healthy Adult Volunteers.
Brief Title: To Evaluate the Pharmacokinetics and the Safety of ID14009 Compared to Coadministration of ID1805 With ID1803 in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-VARE-104
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemias; Hypertension
MeSH Terms: conditions — Dyslipidemias; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ID140009 (Experimental)
  Interventions: Combination Product: ID140009
- ID1803+ID1805 (Active Comparator)
  Interventions: Combination Product: ID1803+ID1805

INTERVENTIONS:
Combination Product: ID140009 — Combination Product: ID140009 Ezetibmibe 10mg/ Rosuvastatin Ca 20.8mg/ Amlodipine 10mg/ Valsartan 160mg
  Arms: ID140009
Combination Product: ID1803+ID1805 — (Amlodipine 10mg/Valsartan 160mg)+(Ezetibmibe 10mg/ Rosuvastatin Ca 20.8mg)
  Arms: ID1803+ID1805

SUMMARY:
To evaluate the pharmacokinetics and the safety of ID14009 compared to coadministration of ID1805 with ID1803 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged over 19 years
* Subjects who have over 50kg and BMI more than 18.5kg/m^2 and less than 29.9kg/m^2
* Subjects who are eligible for this study as determined by clinical laboratory test results, urine test results, vital sign measurements, 12-lead ECG results, and physical examination findings during screening.
* Subjects must agree to practice a medically acceptable method of birth control and should not donate sperm or eggs until 28 days after last dose of study drug.
* Subjects who provided written informed consent to participate in this study and voluntarily taken part in during the entire study period

Exclusion Criteria:

* • Subject with any clinically significant cardiovascular, respiratory, endocrinology, infectious disease, ophthalmology, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease

  * History of gastrointestinal disease (except for appendectomy or herniotomy) or surgery (ex. Crohn's disease, ulcer) that may affect the absorption of a given drug
  * Medical history or evidence that can affect absorption, distribution, metabolism and excretion of a given drug
  * Subject with symptoms of acute disease within 28days prior to study medication dosing
  * Drugs or other drugs (aspirin, antibiotics, etc.) that contain the following drug categories or components of the same strain have an overactive or clinically significant history of hypersensitivity:
  * Subject with a history of drug abuse or urinalysis positive
  * Subject with clinically significant active chronic disease
  * Subject with genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
  * Genetic myopathic disorder or related family history
  * Positive test results for HBs Ab, HCV Ab, Anti HIV(AIDS), RPR Ab
  * Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
  * Subject who cannot take standard meal in hospitalization
  * Present history of hypothyroidism or clinically significant assay
  * Subjects who donated whole blood or partial blood within 2 or 1 month, respectively, prior to the first administration.
  * Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 30days prior to study medication dosing
  * Smokers whose average daily smoking amount exceeds 10 cigarettes per day within 3 months before the first dosing day and those who can't quit from 48 hours before dosing to the time of the last blood sampling.
  * Subjects who judged ineligible by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
AUCt (Total Ezetimibe, Rosuvastatin, Valsartan, Amlodipine) | 0~72hr
  Total Ezetimibe, Rosuvastatin, Valsartan, Amlodipine: AUCt
Cmax (Total Ezetimibe, Rosuvastatin, Valsartan, Amlodipine) | 0~72hr
  Total Ezetimibe, Rosuvastatin, Valsartan, Amlodipine: Cmax

SECONDARY OUTCOMES:
AUCt (Free Ezetimibe) | 0~72hr
  Free Ezetimibe: AUCt
Cmax (Free Ezetimibe) | 0~72hr
  Free Ezetimib: Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- H plus yangji hospital, Seoul, South Korea